CLINICAL TRIAL: NCT02773940
Title: Prospective, Multi-Center Study of the ClariCore™ Optical Biopsy System in Patients Undergoing Radical Retropubic Prostatectomy For Prostate Tissue Classification Algorithm Development
Brief Title: ClariCore™ Biopsy System in Patients Undergoing Radical Retropubic Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Precision Biopsy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STP-1002
Record Dates: First submitted 2016-05-10; First posted 2016-05-16 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ClariCore System (Experimental): Biopsy tissue and correlative spectral data will be acquired using the ClariCore System during the patient's already scheduled radical retropubic prostatectomy (RRP) surgery.
  Interventions: Device: ClariCore System

INTERVENTIONS:
Device: ClariCore System — Biopsy tissue and correlative spectral data will be acquired using the ClariCore System during a patient's already scheduled radical retropubic prostatectomy (RRP) surgery.

SUMMARY:
The purpose of the study is to collect information on prostate tissue biopsies collected with the ClariCore System during a radical prostatectomy procedure. The ClariCore System is designed to improve how biopsies are taken from the prostate by using light sensors (fiber optics) that can see changes in the tissue. The information collected from the study will be used to develop a method to tell the difference between normal and suspicious tissue to help guide the physician during a biopsy procedure.

DETAILED DESCRIPTION:
The overall objective of this study is to acquire and analyze spectral data and correlative tissue biopsy cores using the ClariCore System for the purpose of algorithm development.

The system algorithm will be trained to identify real-time in vivo 'Normal' versus 'Suspicious' prostate tissue. The 'Normal' or 'Suspicious' assignment will be based on the optical signal principle component parameters of the measured signal when compared to a threshold to be derived from pathologically known values of suspicious (or possibly cancerous) and normal (or non-cancerous) measurements in prostate tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for radical retropubic prostatectomy
* Prostate volume > 20cc and height at least 22mm (at the area(s) to be biopsied) as verified by ultrasound or MRI
* Patient, or authorized representative signs a written Informed Consent form to participate in the study, prior to any study mandated determinations or procedure

Exclusion Criteria:

* Patient opted for robotic (da Vinci robot) or laparoscopic surgery
* Any condition, or history of illness or surgery that, in the opinion of the Investigator, might confound the results of the study or pose additional risks to the patient (e.g. significant cardiovascular conditions or allergies)
* Patient has systemic infection or evidence of any surgical site infection (superficial or organ space), including active urinary tract infection
* Bladder cancer (current or prior)
* Actively taking blood thinning agents (with the exception of low dose aspirin {81 mg}, Plavix, Coumadin etc.) or severe medical comorbidity prohibiting halting of anticoagulation therapies or history of bleeding disorder (e.g. coagulopathy)
* Any malignancy other than non-melanoma cell skin cancer, unless no evidence of disease for a minimum of 5 years
* Hormone therapy for locally advanced disease (except patients on 5-alpha reductase inhibitors to reduce the size of the prostate)
* Neo-adjuvant hormonal therapy
* Salvage radical prostatectomy, i.e., patients having surgery due to failure of previous therapy (radiation, brachytherapy, cryotherapy, etc.)
* Patient has compromised immune system or autoimmune disease (WBC < 4000 or > 20,000)
* Patient is not likely to comply with the follow-up evaluation schedule
* Patient is participating in a clinical trial of another investigational drug or device
* Patient is mentally incompetent or a prisoner

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Optical spectra measurements will be correlated with biopsy tissue core samples in patients with known prostate cancer undergoing radical retropubic prostatectomy surgery to develop a prostate tissue classification database | Through study completion which ends at time of procedure completion

SECONDARY OUTCOMES:
All adverse events reported during the procedure that are related to the ClariCore System | Through study completion which ends at time of procedure completion

CONTACTS AND LOCATIONS:
Overall Officials: Alan W Partin, M.D., Ph.D., Principal Investigator — Johns Hopkins University; E. David Crawford, M.D., Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Brady Urological Institute, Johns Hopkins Hospital, Baltimore, Maryland
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No